CLINICAL TRIAL: NCT06585514
Title: Open-Label, Non-Randomized, Single-Arm, Phase 1/2 Study of Anti-CD19 Chimeric Antigen Receptor T Cells for Refractory Systemic Lupus Erythematosus
Brief Title: Anti-CD19 Chimeric Antigen Receptor T Cells for Refractory Systemic Lupus Erythematosus
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing GoBroad Hospital (Other)
Responsible Party: Principal Investigator, Jing Pan, Director of Dept of Hemato-Oncology and Immunotherapy, Beijing GoBroad Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BJGBYY-IIT-LCYJ-2024-040
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2024-11

CONDITIONS: Systemic Lupus Erythematosus (SLE); Lupus Nephritis (LN)
Keywords: Systemic Lupus Erythematosus (SLE); Lupus Nephritis (LN); CD19 CAR-T
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CD19 CAR (Experimental): Following the lymphodepleting treatment, patients will be treated with CD19 Chimeric Antigen Receptor (CAR) positive T cells as a single dose.
  Interventions: Drug: CD19 CAR-T cells

INTERVENTIONS:
Drug: CD19 CAR-T cells — Following lymphodepletion with chemotherapy (cyclophosphamide and fludarabine) patients will be treated with CD19 Chimeric Antigen Receptor (CAR) positive T cells as a single dose.

SUMMARY:
The goal of this study is to evaluate the safety and efficacy of CD19 CAR T cells in the treatment of Systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
This is a single-center, open-label, non-randomized, Phase I/II trial. Patients with refractory systemic lupus erythematosus (SLE) will receive CD19 CAR T cells. The primary objective is to learn about the safety and tolerability of CD19 CAR T cell therapy in subjects with refractory SLE and to determine the optimal biological dose (OBD) and recommend phase 2 dose (RP2D) in phase I and to learn about the efficacy CD19 CAR T-cell therapy in patients with refractory SLE in phase II. The primary endpoint is type and incidence of dose limiting toxicity (DLT) within 28 days after CD19 CAR T-cell infusion in phase I and overall response rate (ORR) in phase II. A total number of 18 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 3-65 years.
2. Have a diagnosis of SLE and meet the classification criteria of 2019 European League Against Rheumatism (EULAR) and the American College of Rheumatology (ACR).
3. Positive antinuclear antibody (ANA): ANA at a titer of ≥ 1:80 on Hep-2 cells or equivalent positive test (ever) and/or a positive anti-dsDNA serum antibody test (based on ELISA assay, ≥ 30 IU/mL).
4. Refractory SLE and/or refractory lupus nephritis (LN):

   • 4.1 Refractory SLE 4.1.1 Patients received at least 7.5 mg/kg/day of prednisolone to maintain low disease activity or the SLEDAI 2K score ≥8.

   4.1.2 Routine treatment is ineffective or the disease relapses after remission. Definition of routine treatment: use glucocorticoid (more than 1mg/kg/d) and cyclophosphamide for 6 months; and any of the following immunomodulatory drugs for more than 3 months: antimalarials, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, and biological agents such as rituximab, belizumab, or telitacicept;

   • 4.2 Refractory LN 4.2.1 Diagnosis of SLE based on the 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR), Biopsy-proven LN class III, IVa [excluding III (C), IV-S (C) and IV-G (C)] or, class V lupus nephritis combined with class III or IV, according to 2018 Revised International Society of Nephrology/Renal Pathology Society (ISN/RPS) criteria, see Appendix 3. Biopsy must be performed within 6 months before or during screening.

   4.2.2 Refractory lupus nephritis is defined as no induced remission to treatment regimens containing at least one immunosuppressant (including glucocorticoids, CTX, tacrolimus, MME, and cyclosporine) after 3 to 6 months, accompanied by no reduction (or worsening) of proteinuria or persistent antibody positives.
5. CD19+ on B cells and continuous withdrawal of the immunosuppressive drugs for more than 1 week.
6. The blood routine lymphocyte count of the subjects is > 1 × 109/L, and there is no cell collection contraindication.
7. No severe allergy.
8. Eastern Cooperative Oncology Group (ECOG) performance status score 0 to 2.
9. Patients are expected to live for at least 90 days.
10. Subjects and/or their guardian must understand and sign the informed consent.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Impaired consciousness or intracranial hypertension:

   * Intracranial pressure elevation was above 15 mmHg;
   * Organic encephalopathy syndrome, cerebrovascular accident, encephalitis or central nervous system vasculitis, visual impairment, and other brain lesions requiring intervention.
2. Symptomatic congestive heart failure or severe cardiac arrhythmia:

   * Previously documented left ventricular ejection fraction (LVEF) by echocardiography of <45% in the 12 months;
   * Abnormal electrocardiogram (ECG): left bundle branch block, bifascicular block or any clinically meaningful ECG abnormality;
   * Congenital long QT syndrome or prolongation of the QT interval corrected for heart rate (QTcF) ≥ 470 ms. QTcF is calculated using Fridericia's Formula;
   * Any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification;
   * Unstable or poorly controlled angina pectoris, including the prinzmetal variant of angina pectoris;
   * Myocardial infarction within 6 months.
3. Manifestations of severe respiratory system failure:

   * Hypoxemic respiratory failure: PaO2 < 60 mmHg, PaCO2 < 50 mmHg at sea level, resting and breathing air conditions;
   * Subjects with pulmonary hypertension (PH): mean pulmonary artery pressure (mPAP) ≥25 mmHg measured by right heart catheterization (RHC);
   * Subjects with hypercapnia (PaCO2 ≥ 50mmHg ) and/or ventilatory dysfunction (PH <7.25 );
   * Oxygen inhalation was required to maintain oxygen saturation;
   * Acute or chronic respiratory diseases unrelated to SLE, such as acute pneumonia and interstitial lung disease.
4. Co-existence with other malignancies.
5. Disseminated intravascular coagulation (DIC).
6. Sepsis or other uncontrollable infections: active uncontrolled systemic bacterial, viral, fungal, or parasitic infection (except for fungal nail infection) or other clinically significant active disease process.
7. Uncontrollable diabetes: after at least 3 months of diet and exercise or similar treatment, fasting blood glucose (FBG) ≥ 8.0 mmol/L, postprandial blood glucose (PBG) ≥ 15 mmol/L, and glycosylated hemoglobin (HbA1c)≥8.0%; diabetic ketoacidosis or other uncontrollable complications of diabetes.
8. Serious mental illness: alcohol or drug abuse, dementia, or any other condition that would impair the subject's ability to receive the planned treatment or to understand informed consent at the study site.
9. Apparent and active intracranial lesions on cranial magnetic resonance imaging (MRI).
10. Underwent organ transplantation, excepting SCT.
11. Pregnant females or lactation.
12. Positive test for infectious hepatitis, acquired immune deficiency syndrome (AIDS) or syphilis.
13. No peripheral blood mononuclear cells (PBMC) collection or frozen PBMC for CAR T cell manufacturing.
14. eGFR CKD-EPI < 30 ml/min/1.73m2.
15. Patients who are unable to discontinue immunosuppression agents for ≥7 days or whose condition recurs during discontinuation while the risk of serious adverse reactions is assessed by the investigator.
16. Any active skin disease that may interfere with the evaluation of SLE, including but not limited to psoriasis, dermatomyositis, systemic sclerosis, non-SLE skin manifestations (e.g., cutaneous vasculopathies, peripapillary dilatation, fingertip sclerosis, rheumatoid nodules, erythema multiforme, leg ulcers), or drug-induced lupus.

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase I: Dose-limiting toxicity (DLT) | 28 days post infusion
  The incidence and type of dose-limiting toxicity (DLT).
Phase I: Adverse events (AEs) | 30 days post infusion
  The incidence and severity of adverse events (AE).
Phase II: Objective response rate (ORR) | 3 months and 6 months post infusion
  Proportions of subjects achieving SLE Responder Index (SRI)-4 response

SECONDARY OUTCOMES:
Phase I: Objective response rate (ORR) | 3 months and 6 months
  Proportions of subjects achieving SLE Responder Index (SRI)-4 response.
Phase I: Long-term Adverse events (AEs) | From 30 days after CD19 CAR T infusion to 2 years
  Total number, incidence and severity of AEs from 30 days to 2 years after CD19 CAR T infusion will be recorded.
Phase I: Pharmacokinetics | Up to 2 years post infusion
  The proliferation and survival of CD19 CAR T cells will be measured by flow cytometry and quantitative polymerase chain reaction (qPCR).
Phase II: Adverse events (AEs) | 2 years post infusion
  The incidence and severity of adverse events.
Phase II: Pharmacokinetics | Up to 2 years post infusion
  The proliferation and survival of CD19 CAR T cells will be measured by flow cytometry and quantitative polymerase chain reaction (qPCR).
Phase II: Overall survival (OS) and during of response (DOR) | Up to 2 years post infusion
  Overall survival (OS) is defined the time from the initial CD19 CAR T cell infusion to death for any cause. During of response (DOR) is defined as the date when response criteria are first met to the date of relapse or death caused by SLE in the absence of documented relapse.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing GoBroad Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Results will be published anonymized and summarized.